CLINICAL TRIAL: NCT06166693
Title: A Randomized Controlled Trial of a Personality Trait-focused Digital Mental Health Intervention
Brief Title: The Effectiveness of the "MINDLiNG" Digital Mental Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 40FY (Industry)
Collaborators: The Ministry of SMEs and Startups. South Korea (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SNUH_MINDLiNG_RCT
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Mental Health Services; Personality
Keywords: digital mental health service; intervention; randomized controlled trial; Personality Focused

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Adults between the ages of 18 and 60 were recruited and randomly assigned to the treatment group and waitlist group in the ratio of 2:1. Based on the screening results, 75 participants were assigned to each of the four intervention programs within MINDLiNG (Riggy, Pleaser, Shelly, and Jumpy).
  Interventions: Device: "MINDLiNG" Digital Mental Health Intervention
- Waitlist group (No Intervention): Adults between the ages of 18 and 60 were recruited and randomly assigned to the treatment group and waitlist group in the ratio of 2:1. Based on the screening results, 25 participants were assigned to each of the four intervention programs waitlist.

INTERVENTIONS:
Device: "MINDLiNG" Digital Mental Health Intervention — The intervention was delivered on an online platform set up separately for the study, which was accessible via the web browser and application. The psychological intervention program for maladaptive personality traits (Mindling) is based on the principles of CBT, psychological schema therapy, acceptance-commitment therapy, and mindfulness-based cognitive therapy, and is aimed primarily at adults to prevent and overcome psychological difficulties
  Arms: Treatment group

SUMMARY:
A study in South Korea assessed the effectiveness of the "MINDLiNG" digital mental healthcare program, targeting maladaptive personality traits, and found significant improvements in reducing stress, perfectionism, loneliness, and anxiety, while increasing self-esteem among participants. The study highlights the potential of digital solutions to address the high demand for mental healthcare services in South Korea.

DETAILED DESCRIPTION:
This study conducted a randomized controlled trial to evaluate the effectiveness of a digital intervention program called "MINDLiNG" designed to target maladaptive personality traits, with four subprograms addressing perfectionism, low self-esteem, social isolation, and anxiety. Participants were assigned to one of these programs, and primary outcome measures varied accordingly, including the Perceived Stress Scale, Hewitt Multidimensional Perfectionism Scale, State Self-Esteem Scale, UCLA Loneliness Scale, and Beck Anxiety Inventory. The study anticipated treatment effects in both primary and secondary outcome measures for the treatment group compared to the waitlist group after 5 and 10 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 60
* Experiencing a moderate level of stress in their daily lives (PSS≥17) and meet a certain level of perfectionism (HMPS≥198), self-esteem (SSES≤57), loneliness (UCLA LS≥47), and anxiety (BAI≥16). The cutoff points for each scale are based on the top or bottom 25% of the frequency distribution suggested in the previous study.

Exclusion Criteria:

* In cases where there is difficulty understanding and reading Korean.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | The treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  The primary outcome measure for the entirety of the MINDLiNG program. The Perceived Stress Scale (PSS) is a 10-item scale that can range from 0 to 40, which measures the perceived stress on a 5-point severity with higher scores indicating more severe perceived stress.
Hewitt Multidimensional Perfectionism Scale | The Riggy treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  Perfectionism, the primary outcome of the Riggy program, was measured using the Hewitt Multidimensional Perfectionism Scale (HMPS).
  The HMPS is a 45-item measure with three trait subscales measuring self-oriented perfectionism, other-oriented perfectionism, and socially prescribed perfectionism. It ranges from 45 to 315. Higher level means higher level of perfectionism.
State Self-Esteem Scale | The Pleaser treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  State self-esteem, the primary outcome of the Pleaser program, was measured using the Sate Self-Esteem Scale (SSES) SSES is a 20-item scale on a 5-point likert scale ranging from 20 to 100, assessing 3 facets of self-esteem: appearance, performance, and social. Higher score means higher level of self-esteem.
UCLA Loneliness Scale | The Shelly treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  Loneliness, the primary outcome of the Shelly program, was measured using the UCLA Loneliness Scale (UCLA-LS).
  UCLA-LS is a 20-item scale to measure subjective feelings of loneliness as well as feelings of social isolation on a 4-point likert scale ranging from 20 to 80. Higher score means higher level of loneliness.
Beck Anxiety Inventory (BAI) | The Jumpy treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  The primary measure of the Jumpy program was the BAI. A 21-item self-inventory on a 4-point likert scale ranging from 0 to 63, measuring common somatic and cognitive symptoms of anxiety. Higher score means higher level of anxiety

SECONDARY OUTCOMES:
Self-Efficacy Stress (SES) | The treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  A measure for entirety of the MINDLiNG program. The SES is a 23-item scale that assesses the individuals self-efficacy on a 5-point likert scale ranging from 23 to 115. Higher scores indicate higher level of self-efficacy.
Center for Epidemiologic Studies Depression Scale (CES-D) | The treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  A measure for entirety of the MINDLiNG program. The CES-D is a 20-item questionnaire that measures depressive symptoms on a 4-point likert scale ranging from 0 to 60. Higher score means higher level of depression.
State-Trait Anxiety Inventory (STAI) trait | The treatment group was assessed at Weeks 0, 5, 10, and 14, and the waitlist group at Weeks 0, 5, and 10
  A measure for entirety of the MINDLiNG program. The STAI trait is a 20-item inventory that measures trait anxiety on a 4-point likert scale ranging from 20 to 80. Higher score means higher anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Sup Shin, PhD, Principal Investigator — Seoul National University College of Medicine, Department of Psychiatry
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeong S, Kim H, Lho SK, Hwang I, Mun S, Kim S, Lim H, Kim H, Shin MS, Moon W. Schema-Informed Digital Mental Health Intervention for Maladaptive Cognitive-Emotional Patterns: Randomized Controlled Trial. J Med Internet Res. 2025 Aug 14;27:e65892. doi: 10.2196/65892. PMID 40574385